CLINICAL TRIAL: NCT06872996
Title: Trophallergen Prick Tests (PT) : Influence of Food Sample Shelf Life on the Reproducibility of PT Results
Acronym: TROPHAPRICK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUO-2024-19
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Food Allergy
Keywords: Prick test; Skin test; Trophallergen; Food sample; Fresh; Frozen; Fruit; vegetables; Meat; Alpha-gal; Arachide; Leguminous plant; Milk; Nuts; Fish; Seafood
MeSH Terms: conditions — Food Hypersensitivity | interventions — Patch Tests

STUDY DESIGN:
Intervention Model Description: Participants are recruited, day by day, according to the modalities and eligibility criteria during consultations or day hospitalizations in the allergology department of Orléans University Hospital for the follow-up of their food allergy.
  All participants present one or more food allergy(ies) followed at Orléans University Hospital and agree to participate in the TROPHAPRICK study.
  If a potential patient attends a consultation without their native foods, the investigator will not include them in the study. However, they may participate in the study during a subsequent follow-up consultation with the investigator (if recruitment is still ongoing).
  The duration of the inclusion period is maximum 30 months (upon inclusion of the 100th patient) Each participant follow-up duration is 30 minutes (maximum 1 hour) The total research duration is 30 months maximum. The end of the study is defined as the date of the last visit of the last patient.
Masking Description: In the context of the study, one person will perform the PT, and a second person, blinded, will read the tests. This second person will not know the order of the PT performed (fresh food versus preserved food).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Food allergies arm (Experimental): The participants are their own control. Performing all tests in a single session avoid analysis biases related to intra-individual variability in reactivity encountered during prick-tests performed on various dates (patient included only once in the study, no possible re-inclusion).
  Interventions: Diagnostic Test: Prick-test

INTERVENTIONS:
Diagnostic Test: Prick-test — Several foods may be tested for the same participant depending on the number of food allergies the patient has. PT are performed using the "prick-to-prick" method with lancets, in a single session per patient, using fresh and preserved native foods. Simultaneously, a positive control and a negative control are performed. The PT are performed and read by nursing or medical staff trained in the technique.
  Participants' clinical follow-up is performed continuously for 30 minutes from the performance of the prick-tests and under the responsibility of the allergologist doctor, whose presence is mandatory during the performance of these tests.
  For meat, fruit, vegetable, leguminous plant, milk, seafood and fish tests will be performed with fresh products and with products preserved for 3 months as well as with products preserved for 6 months [-15 days; +15 days].
  For dry foods (nuts and peanuts), tests will be performed with products harvested over 3 separate and consecutive seasons.

SUMMARY:
Prick tests (PT) are the standard skin tests used in the investigation of immediate IgE-mediated food allergies. Their use as a first-line tool in allergological investigations is strongly recommended by the European Academy of Allergy and Clinical Immunology (EAACI). These tests involve locally reproducing histamine release manifestations in the epidermis by superficially introducing an allergen to confirm or rule out its role in the onset of clinical symptoms compatible with an allergy. During the diagnostic management and follow-up of patients with food allergies, the technique used is the "prick to prick" method, due to the lack of reliable access to many standardized commercial food extracts. This method involves piercing the food with a sterile lancet (to deposit food content on its surface) and then making a superficial skin puncture with the same device on the anterior surface of the forearm to introduce a tiny fraction of the food and its proteins into the epidermis, where mast cells are present. Simultaneously, a positive control and a negative control are performed. The tests are read after 15 to 20 minutes by measuring the size in millimeters of the resulting papules and erythema. A PT for the tested allergen is considered positive if the average diameter of the resulting papule is 3 mm or more and/or at least half the size of the positive control papule. The procedure is well-tolerated, allowing it to be performed at any age, in both hospital and outpatient settings. The risk of a systemic reaction has been evaluated at 0.008%, with no severe reactions observed.

This method, performed with native foods (unprocessed food, uncontaminated foods), either raw or cooked (depending on the nature of the allergen being tested), is preferred over the use of commercial extracts (standardized commercial allergen preparations) due to its better sensitivity and specificity, the high cost of commercial extracts, and the lack of commercial extracts for certain foods. For practical reasons, given the wide variety of possible allergens, and to most accurately reproduce the exposure that caused the reaction, the most common approach is to ask the patient to bring their own foods for testing. These foods should be brought in a fresh state. However, situations where the patient is offered a food PT but does not have fresh native foods are common. Indeed, many patients forget to bring them. Similarly, during a consultation to explore a respiratory or drug allergy, the interview may lead to the detection of a food allergy that needs to be tested at the same time. Given the delays in allergology consultations, the severity of food allergy symptoms, and the potential risk of delayed diagnosis, all allergists involved in managing food allergies are led to create a library of food samples stored either in a dry state (e.g., nuts, peanuts, cereal flours) or frozen for perishable foods (meats, shellfish, fruits, vegetables). To our knowledge, after reviewing the literature, no guidelines for best practices regarding the storage of these food samples for PT purposes have been established by scientific societies. Moreover, while the impact of freezing and thawing methods on the denaturation of food proteins is known, the effect of freezing and its duration on the sensitivity and specificity of PT is poorly understood.

The objective of our study is to evaluate the reproducibility of PT results between those performed with fresh foods and those performed with preserved foods at different storage dates in participants who have experienced anaphylaxis of at least grade 2 according to the Ring and Messmer classification.

DETAILED DESCRIPTION:
Interventional, exploratory, prospective, single-center clinical study comparing for each patient included, at the same time, the results of prick tests carried out with fresh native food allergens and those carried out with native foods stored for prolonged period (in the freezer or dry dependig on the nature of the product) and for different shelf lives.

A native food is a raw food not contaminated by other foods. It is said to be fresh if it has not been subject to a prolonged preservation technique such as freezing or canning. The native food can be raw or cooked depending on the nature of the food and the nature of the allergic protein tested.

In our study the patient is his own witness. Carrying out all tests in a single session makes it possible to avoid analysis biases related to intra-individual variabilities in reactivity encountered during prick tests carried out on different dates (patient included only once in the study, no re-inclusion possible). In our study, several foods can be tested for the same patient depending on the number of food allergies that the patient has.

The completion of the study does not change the follow up methods for patients who are already offered prick tests as part of their allergic pathology. The study lasts approximately 30 minutes for each patient, while the prick tests are carried out. Their follow up is carried out by nurses of the allergology department for 30 minutes from the completion of the prick tests and this, under the responsibility of the allergist doctor of the department whose presence is obligatory when performing these tests.

Participants will be fully and honestly informed, in understandable terms, about the objectives and constraints of the study, the potential risks incurred, the necessary monitoring and safety measures, and their rights to refuse to participate in the study or to withdraw at any time.

All this information is provided in an information form given to the patient. The patient's written consent will be obtained by the investigator, a junior doctor, or a representative doctor before any procedure specific to the study.

As this is a pilot, exploratory, monocentric study, and given that Orléans University Hospital receives approximately 50 patients per year (who meet the eligibility criteria), it is planned to include 100 patients in the study over a maximum period of 30 months.

A clinical research associate (ARC) mandated by the sponsor will ensure the proper conduct of the study, the collection of generated data, its documentation, recording, and reporting, in accordance with the Standard Operating Procedures implemented within Orléans University Hospital and in compliance with Good Clinical Practices as well as the applicable legislative and regulatory provisions.

Participants will be fully and honestly informed, in understandable terms, about the objectives and constraints of the study, the potential risks incurred, the necessary monitoring and safety measures, and their rights to refuse to participate in the study or to withdraw at any time.

All this information is provided in an information form given to the patient. The patient's written consent will be obtained by the investigator, a junior doctor, or a representative doctor before any procedure specific to the study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and over.
2. Having a diagnosis of food allergy(ies) due to one or more of the food allergen studied, previously made by an allergologist, of grade 2 to 3 according to the Ring and Messmer classification.
3. Having given consent to participate in the study.

The diagnosis is made by the allergologist of the department due to the presence of a compatible clinical history implicating the tested allergen, the presence of evidence of sensitization to the allergen (positive prick-test and/or positive specific IgE assays), or even a positive oral allergen reintroduction test.

Exclusion Criteria:

1. Anaphylactic reaction dating less than 6 weeks
2. Hospitalization for asthma in the past 3 months
3. History of grade 4 anaphylactic reaction according to the Ring and Messmer classification.
4. Systemic antihistamine treatment in the 7 days preceding the test
5. Systemic beta-blocker treatment on the day of the test.
6. Protected person (under guardianship or curatorship)
7. Person under judicial supervision
8. Persons deprived of liberty
9. Person not affiliated with a social security insurance
10. Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-10-10 (Estimated); Study Completion 2027-10-10 (Estimated)

PRIMARY OUTCOMES:
Average diameter (mm) of the resulting papules obtained from PT performed with fresh foods, with preserved foods at different storage durations and with positives and negatives controls. | The tests are read 15 to 20 minutes after the food is pricked onto the participants' skin
  Average diameter of the papule : average between the smallest diameter and the largest diameter of the papule.
  Test interpretable if the average diameter of the positive histamine control papule is 3 mm or more and if the average diameter of the negative saline control papule is less than 3 mm.
  Test considered positive if the average diameter of the papule obtained with the allergen is 3 mm or more and/or half or more of the size of the positive control papule.
  Test considered negative if the average diameter of the papule obtained with the allergen is less than 3 mm.

SECONDARY OUTCOMES:
The Histamine Equivalent Prick index diameter (HEP-index diameter) calculated during PT performed with fresh foods and foods stored for different durations | The tests are read 15 to 20 minutes after the food is pricked onto the participants' skin.
  The HEP-index diameter (Histamine Equivalent Prick index diameter) obtained by dividing the average diameter of the papule induced by the allergen by the average diameter of the positive histamine control papule.
  Test interpretable if the average diameter of the positive histamine control papule is 3 mm or more and if the average diameter of the negative saline control papule is less than 3 mm.
  Test considered positive if HEP-index diameter is 0.6 or more. Test considered negative if HEP-index diameter is less than 0.6.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire d'Orléans, Orléans, France

REFERENCES:
- [Background] Santos AF, Riggioni C, Agache I, Akdis CA, Akdis M, Alvarez-Perea A, Alvaro-Lozano M, Ballmer-Weber B, Barni S, Beyer K, Bindslev-Jensen C, Brough HA, Buyuktiryaki B, Chu D, Del Giacco S, Dunn-Galvin A, Eberlein B, Ebisawa M, Eigenmann P, Eiwegger T, Feeney M, Fernandez-Rivas M, Fisher HR, Fleischer DM, Giovannini M, Gray C, Hoffmann-Sommergruber K, Halken S, Hourihane JO, Jones CJ, Jutel M, Knol E, Konstantinou GN, Lack G, Lau S, Marques Mejias A, Marchisotto MJ, Meyer R, Mortz CG, Moya B, Muraro A, Nilsson C, Lopes de Oliveira LC, O'Mahony L, Papadopoulos NG, Perrett K, Peters RL, Podesta M, Poulsen LK, Roberts G, Sampson HA, Schwarze J, Smith P, Tham EH, Untersmayr E, Van Ree R, Venter C, Vickery BP, Vlieg-Boerstra B, Werfel T, Worm M, Du Toit G, Skypala I. EAACI guidelines on the diagnosis of IgE-mediated food allergy. Allergy. 2023 Dec;78(12):3057-3076. doi: 10.1111/all.15902. Epub 2023 Oct 10. PMID 37815205
- [Background] Riggioni C, Ricci C, Moya B, Wong D, van Goor E, Bartha I, Buyuktiryaki B, Giovannini M, Jayasinghe S, Jaumdally H, Marques-Mejias A, Piletta-Zanin A, Berbenyuk A, Andreeva M, Levina D, Iakovleva E, Roberts G, Chu D, Peters R, du Toit G, Skypala I, Santos AF. Systematic review and meta-analyses on the accuracy of diagnostic tests for IgE-mediated food allergy. Allergy. 2024 Feb;79(2):324-352. doi: 10.1111/all.15939. Epub 2023 Nov 27. PMID 38009299
- [Background] Henzgen M, Ballmer-Weber BK, Erdmann S, Fuchs T, Kleine-Tebbe J, Lepp U, Niggemann B, Raithel M, Reese I, Saloga J, Vieths S, Zuberbier T, Werfel T; German Society of Allergology and Clinical Immunology (DGAKI); Physicians' Association of German Allergologists (ADA); Society of Pediatric Allergology (GPA); Swiss Society of Allergology. Skin testing with food allergens. Guideline of the German Society of Allergology and Clinical Immunology (DGAKI), the Physicians' Association of German Allergologists (ADA) and the Society of Pediatric Allergology (GPA) together with the Swiss Society of Allergology. J Dtsch Dermatol Ges. 2008 Nov;6(11):983-8. doi: 10.1111/j.1610-0387.2008.06889.x. English, German. PMID 18992038
- [Background] Rance F, Juchet A, Bremont F, Dutau G. Correlations between skin prick tests using commercial extracts and fresh foods, specific IgE, and food challenges. Allergy. 1997 Oct;52(10):1031-5. doi: 10.1111/j.1398-9995.1997.tb02427.x. PMID 9360758
- [Background] Brockow K, Romano A, Blanca M, Ring J, Pichler W, Demoly P. General considerations for skin test procedures in the diagnosis of drug hypersensitivity. Allergy. 2002 Jan;57(1):45-51. No abstract available. PMID 11991289
- [Background] Ruethers T, Johnston EB, Karnaneedi S, Nie S, Nugraha R, Taki AC, Kamath SD, Williamson NA, Mehr SS, Campbell DE, Lopata AL. Commercial shellfish skin prick test extracts show critical variability in allergen repertoire. Allergy. 2023 Dec;78(12):3261-3265. doi: 10.1111/all.15853. Epub 2023 Aug 21. No abstract available. PMID 37602511
- [Background] Patti ML, De Rose C, Brancato F, Gambacorta A, Miceli Sopo S. Sensitivity of prick test with walnut commercial extracts and of prick by prick with raw walnut compared with open food challenge in walnut allergy. Acta Biomed. 2021 Apr 30;92(S1):e2021067. doi: 10.23750/abm.v92iS1.10043. PMID 33944826
- [Background] Codreanu F, Moneret-Vautrin DA, Morisset M, Guenard L, Rance F, Kanny G, Lemerdy P. The risk of systemic reactions to skin prick-tests using food allergens: CICBAA data and literature review. Eur Ann Allergy Clin Immunol. 2006 Feb;38(2):52-4. PMID 16711536
- [Background] Lee S, Jo K, Jeong HG, Choi YS, Kyoung H, Jung S. Freezing-induced denaturation of myofibrillar proteins in frozen meat. Crit Rev Food Sci Nutr. 2024;64(5):1385-1402. doi: 10.1080/10408398.2022.2116557. Epub 2022 Sep 2. PMID 36052640
- [Background] Garriga T, Guilarte M, Luengo O, Guillen M, Labrador-Horrillo M, Fadeeva T, Sala A, Cardona V. Frozen fruit skin prick test for the diagnosis of fruit allergy. Asian Pac J Allergy Immunol. 2010 Dec;28(4):275-8. PMID 21337912
- [Background] Terlouw S, van Boven FE, Borsboom-van Zonneveld M, de Graaf-In 't Veld T, Gerth van Wijk R, van Daele PLA, van Maaren MS, Kuijpers JHSAM, Veenbergen S, de Jong NW. Comparison of skin prick test and prick-to-prick test with fruits and vegetables in the diagnosis of food allergy. Clin Transl Allergy. 2024 Jul;14(7):e12375. doi: 10.1002/clt2.12375. PMID 38970153
- [Background] Begin P, Des Roches A, Nguyen M, Masse MS, Paradis J, Paradis L. Freezing does not alter antigenic properties of fresh fruits for skin testing in patients with birch tree pollen-induced oral allergy syndrome. J Allergy Clin Immunol. 2011 Jun;127(6):1624-6.e3. doi: 10.1016/j.jaci.2011.01.028. Epub 2011 Mar 16. No abstract available. PMID 21411128
- [Background] van der Valk JP, Gerth van Wijk R, Hoorn E, Groenendijk L, Groenendijk IM, de Jong NW. Measurement and interpretation of skin prick test results. Clin Transl Allergy. 2016 Feb 23;6:8. doi: 10.1186/s13601-016-0092-0. eCollection 2015. PMID 26909142
- [Background] Warren CM, Sehgal S, Sicherer SH, Gupta RS. Epidemiology and the Growing Epidemic of Food Allergy in Children and Adults Across the Globe. Curr Allergy Asthma Rep. 2024 Mar;24(3):95-106. doi: 10.1007/s11882-023-01120-y. Epub 2024 Jan 12. PMID 38214821
- [Background] Dribin TE, Motosue MS, Campbell RL. Overview of Allergy and Anaphylaxis. Emerg Med Clin North Am. 2022 Feb;40(1):1-17. doi: 10.1016/j.emc.2021.08.007. Epub 2021 Oct 29. PMID 34782082
- [Background] Pax AP, Ong L, Pax RA, Vongsvivut J, Tobin MJ, Kentish SE, Gras SL. Industrial freezing and tempering for optimal functional properties in thawed Mozzarella cheese. Food Chem. 2023 Mar 30;405(Pt B):134933. doi: 10.1016/j.foodchem.2022.134933. Epub 2022 Nov 12. PMID 36410214
- [Background] Bao Y, Ertbjerg P, Estevez M, Yuan L, Gao R. Freezing of meat and aquatic food: Underlying mechanisms and implications on protein oxidation. Compr Rev Food Sci Food Saf. 2021 Nov;20(6):5548-5569. doi: 10.1111/1541-4337.12841. Epub 2021 Sep 25. PMID 34564951